CLINICAL TRIAL: NCT03990064
Title: Exploration of Cerebral Metabolism and Connectivity in Post Traumatic Stress Disorder (PTSD): Exploratory Study of Neurofunctional Modulation of Emotions by Music Therapy
Brief Title: Benefits of Relaxation by Music Therapy on PTSD Symptoms
Acronym: TRACER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Principal Investigator, Marion Trousselard, principal investigator, Institut de Recherche Biomedicale des Armees
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-A02182-53
Record Dates: First submitted 2019-05-08; First posted 2019-06-18 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Stress Disorder, Post Traumatic
Keywords: effective connectomic neurological soft signs
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: musicotherapy versus waiting list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- musicotherapy (Experimental): daily sessions of music listening during 2 months, associated with their standard treatment,
  Interventions: Other: musicotherapy
- waiting list (No Intervention): waiting list

INTERVENTIONS:
Other: musicotherapy — receptive music therapy. The musical style of the session was chosen by the patient. The validated 'U' technique was employed.
  Arms: musicotherapy

SUMMARY:
PTSD is a debilitating mental disorder that may develop after experiencing or witnessing a life-threatening event. With appropriate care, treatment efficiency is variable and around 20% of the patients do not respond to psychological treatment. Complementary treatments are needed.

as PTSD implied autonomic nervous system (ANS) dysfonction, complementary treatment focusing on ANS regulation, as welle as musicotherapy, may have an interest.

DETAILED DESCRIPTION:
The aim is to evaluate the impact of musicotherapy on PTSD symptoms, and severity using a RCT Symptoms will be evaluated using questionaires (PCL and quality of life) severity will be measured using neurological soft signs assessment, connectomic functions and ANS regulation

ELIGIBILITY:
Inclusion Criteria:

* PTSD

Exclusion Criteria:

* neurological diseases
* addiction

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
change in PTSD symptoms | change from PTSD symptoms at two months and at six months
  questionnaire Posttraumatic CheckList 5 (PCL5; threshold =33)

SECONDARY OUTCOMES:
change in neurological soft signs | change from neurological soft signs at two months and at six months
  questionnaire EPSID " Psychomotor assessment scale of neurological soft signs no threshold
change in effective connectomic | change from effective connectomic at two months and at six months
  Magnetic Resonance Imaging
Autonomous nervous system regulation | change from Autonomous nervous system regulation at two months and at six months
  heart rate variability during 5 min at rest
change in biological stress | change from biological stress at two months and at six months
  blood cytokines, BDNF

CONTACTS AND LOCATIONS:
Locations (1):
- Marion TROUSSELARD, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No